CLINICAL TRIAL: NCT05043753
Title: Department of Obstetrics and Gynecology Modena Policlinico Hospital Vial Del Pozzo 71, 41125 Modena
Brief Title: "Fetal GRowth AbnorMality DEtection Trial"
Acronym: FRAME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Giuseppe Chiossi, Attending Physician, Department of Obstetrics and Gynecology, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: University of Modena
Record Dates: First submitted 2021-09-02; First posted 2021-09-14 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Small for Gestational Age Infant; Large for Gestational Age Infant; Oligohydramnios; Polyhydramnios
MeSH Terms: conditions — Oligohydramnios; Polyhydramnios

STUDY DESIGN:
Intervention Model Description: To compare the diagnostic accuracy of symphysis fundal height (SFH) as opposed to SFH combined with point of care ultrasound to measure the fetal abdominal circumference (POC-US-AC) in identifying small and large for gestational age infants (SGA and LGA infants) among low-risk pregnant women cared for by midwives after 35 weeks' gestation.
  Low risk pregnancies will be evaluated at 35-38, 40, 41, and 41+ weeks' gestation by midwives trained in SFH measurement and POC-US. Formal obstetric US performed by a perinatologist (i.e high risk obstetrician) will be performed in case SFH and/or POC-US suspect fetal growth or amniotic fluid abnormalities. Prenatal evaluations will be compared to actual birthweights
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group: Symphysis fundal height measurement (No Intervention): Screening for fetal growth abnormalities is performed by certified nurse midwives (CNMs) using symphysis fundal height (SFH)
- intervention group: Symphysis fundal height measurement and point of care ultrasound. (Experimental): Screening for fetal growth abnormalities is performed by certified nurse midwives (CNM) using symphysis fundal height (SFH) and point of care ultrasound to measure the fetal abdominal circumference (POC-US-AC)
  Interventions: Other: Point of care ultrasound to measure the fetal abdominal circumference (POC-US-AC)

INTERVENTIONS:
Other: Point of care ultrasound to measure the fetal abdominal circumference (POC-US-AC) — Midwives perform a POC-US to measure the fetal abdominal circumference (AC) and evaluate the quantity of amniotic fluid.
  In order to identify the appropriate sonographic plane the following markers need to be identified on POC-US
  * Fluid filled fetal stomach on the left.
  * Umbilical vein
  * Umbilical portion of left portal vein within liver, as it meets the "pars transversa" (horizontal portion of left portal vein) seen as a right sided " L " or " C " shape.
  * Fetal spine seen in cross section Amniotic fluid volume will be evaluated determining the deepest vertical pocket (DVP). Measurement is performed by assessing a pocket of maximal depth of amniotic fluid free of umbilical cord and fetal parts. The transducer is held perpendicularly to the patient's abdomen. The absence of a pocket measuring at least 2 cm in depth and 1 cm in width is indicative of oligohydramnios, while detection of a pocket measuring 8 cm or larger is suggestive of polyhydramnios (ACOG bulletin 175, 2016).
  Other Names: Bedside ultrasound
  Arms: intervention group: Symphysis fundal height measurement and point of care ultrasound.

SUMMARY:
The present trial intends to assess the diagnostic accuracy of symphysis fundal height (SFH) as opposed to SFH combined with point of care ultrasound to measure the fetal abdominal circumference (POC-US-AC) in identifying small and large for gestational age infants (SGA and LGA infants) among low-risk pregnant women cared for by midwives after 35 weeks' gestation.

Low risk pregnancies will be evaluated at 35-38, 40, 41, and 41+ weeks' gestation by midwives trained in SFH measurement and POC-US. Formal obstetric US performed by a perinatologist (i.e high risk obstetrician) will be performed in case SFH and/or POC-US suspect fetal growth or amniotic fluid abnormalities. Prenatal evaluations will be compared to actual birthweights.

DETAILED DESCRIPTION:
Birthweight below the 10th (small for gestational age or SGA) or above the 90th (large for gestational age or LGA) percentile for gestational age has been associated with adverse maternal, fetal and neonatal outcomes. As birthweight reflects intrauterine development, accurate identification of abnormal fetal growth would allow obstetric providers to prevent adverse outcomes and mitigate complications associated with abnormal development.

Symphysis fundal height (SFH) measured in centimeters after 24 weeks of gestation is recommended as the standard of care to screen for fetal growth abnormalities among low-risk pregnancies. This method is low-cost, and easy to perform, but there is a lack of evidence supporting its effectiveness due to its poor sensitivity. Ultrasonography, the technique utilized to identify fetal growth abnormalities, is a costly procedure which involves the use of advanced equipment and providers, to perform and review the ultrasound, as well as a full examination with multiple measurements and images. Despite a few encouraging reports, insufficient evidence supports routine 3rd trimester ultrasound in low- risk pregnancies to improve detection of abnormal fetal growth.

Sonographic measurement of the abdominal circumference (AC) in the fetus was shown to be the single most useful indicator of fetal growth. Measurement of AC does not require extensive training, long time to acquire, or expensive ultrasound machines. It can be easily performed in the office by midwives who are specifically trained in obtaining the measurement. Therefore, we intended to evaluate if the use of bedside point of care ultrasound (POC-US) by midwives to evaluate fetal AC during routine antenatal visits in low-risk pregnancies would increase the accuracy of SFH in identifying fetuses with birthweight < 10th or > 90th, when compared to SFH alone.

This is an open label, investigator sponsored, two arms randomized controlled trial. Patients who satisfy all inclusion criteria, have no exclusion criteria, and have signed the written informed consent will be randomly assigned to screening of fetal growth abnormalities during routine antenatal appointments held by midwives according to SFH or SFH + POC-US-AC.

Low risk pregnant women are interviewed by a midwife at 35-38 weeks' gestation, who also reviews their medical and obstetrical history, prenatal labs and the ultrasound reports to discriminate between high and low-risk pregnancies. Patients who satisfy all inclusion criteria and do not have any exclusion criteria will be randomly assigned to one of two different approaches to identify fetal growth abnormalities and predict abnormal birthweight, after signing the written informed consent.

Screening test in the control group: Symphysis fundal height measurement. Fundal height is measured by trained midwives at each scheduled antenatal appointment from the pubis symphysis to the top of the uterine fundus, using a paper measuring tape in centimeters. Size greater than dates is suspected if the measurement is above the 90th gestational age specific percentile according to the Intergrowth 21 SFH references (Papageorghiu 2016). Similarly, size less than dates is recorded if the measurement is below the 10th percentile for age according to the Intergrowth 21 SFH references (Papageorghiu 2016). Formal obstetric ultrasound is requested if the SFH is > 90th percentile, if it is < 10th , or if it drops 50 growth centiles in two subsequent evaluations.

Screening test in the intervention group: Symphysis fundal height measurement + point of care ultrasound. After assessing SFH at each clinical encounter, the midwife will perform a POC-US to measure the fetal AC and evaluate the quantity of amniotic fluid. A positive screen for fetal growth restriction (indicative of a potential SGA infant) consists in a measured AC less than the 10th percentile for gestational age according to the standards defined by Nicolini et al in 1986 on an Italian population; instead, a positive screen for macrosomia (suggestive of a potential LGA infant) is an AC greater than the 90th percentile for gestational age according to the references set by Nicolini et al in 1996. Formal obstetric ultrasound is requested if the AC is > 90th percentile, if it is < 10th, or if it drops 50 growth centiles in two subsequent evaluations. Amniotic fluid volume will be evaluated determining the deepest vertical pocket (DVP).

A formal US is requested in case uterine size is measured as ≤ than the 10th or ≥ than the 90th percentile for gestational age according to Intergrowth 21, when POC - US reveals AC < 10th percentile, AC > 90th percentile according to Nicolini et al, in case DVP < 2 x 1 cm, or DVP > 8 x 1 cm, or also if SFH or AC drop > 50 percentiles comparing two subsequent evaluations. Patients randomized to SFH + POC-US will have a formal US if either technique suspects abnormal fetal growth.

Formal US requested due to an abnormal screening test will be distinguished from scans ordered due to other indications, such as hypertensive disorders of pregnancy, or cholestasis of pregnancy diagnosed after enrollment. Hadlock' s references will be used to estimate fetal weight, and therefore to define FGR (i.e estimated fetal weight or AC < 10th percentile) as well as macrosomia (i.e estimated fetal weight or AC > 90th percentile).

Prenatal evaluation of fetal growth will be compared to the birthweight percentile according to the INeS neonatal charts (Bertino 2010) to identify SGA, LGA and AGA (appropriate for gestational age) infants.

After the initial evaluation low risk pregnancies are scheduled for antenatal appointments with a midwife at 40, 41 and 41+ weeks' gestation. All patients will have a POC-US by a midwife at 41, and 41+ weeks' gestation to screen for amniotic fluid abnormalities associated with protracted pregnancy, independently of the randomization arm. A midwife will perform SFH or SFH + POCT-US (according to randomization) at enrolment (35-38 weeks' gestation) and at 40 weeks. As sonographic assessment of fetal growth should not be performed more frequently than every 2 weeks due to the error associated with measurements; POC-US will only evaluate amniotic fluid volume at 41 and 41+3 weeks' gestation (unless the patient has missed a previous appointment), even among women randomized to SFH + POC-US.

The purpose of the study is to evaluate the most accurate approach to identify prenatally those pregnancies that will result in SGA or LGA infants. Prenatal evaluation consists in a universal screening test for fetal growth abnormalities (either SFH or SFH + POC US) followed by a confirmatory test (formal obstetric US) performed only when the initial screening test is positive. Fetal growth or amniotic fluid abnormalities are diagnosed in utero if confirmed by a formal obstetric ultrasound, and not when only suspected by a screening test; in fact, the study seeks to evaluate what is the most accurate combination of screening and confirmatory tests, and not the effectiveness of the screening test alone.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥ 18 years and ability to give informed consent.
* Singleton gestation
* Ultrasound examination that confirms or revises the EDD before 14 weeks of gestational age
* Gestational age ≥ 35 weeks' gestation
* Normal aneuploidy screening (1st trimester screening, 2nd trimester screening, integrated screening, NIPT) when performed
* Spontaneously conceived pregnancy (i.e the current pregnancy is not the result of in vitro fertilization)

Exclusion Criteria:

* Fetal chromosomal or genetic abnormalities if invasive prenatal diagnosis is performed
* Fetal malformations or soft markers identified on fetal anatomy survey
* Episodes of uterine bleeding after 24 weeks gestation. Unobserved self-reported bleeding with confirmed intact pregnancy on ultrasound after the bleeding episode is not an exclusion criteria.
* Uterine/placental abnormalities including uterine malformations (i.e bicornuate uterus, didelpus uterus), abnormal placentation (placenta previa, accreta, percreta), uterine fibroids.
* Cerclage in the current pregnancy
* History of intrauterine fetal demise
* History of fetal growth restriction or birth weight > 4Kg in a previous pregnancy
* Fetal isoimmunization or alloimmunization
* Fetal demise in previous pregnancies
* Cancer (including melanoma but excluding other skin cancers). Dysplastic or pre-neoplatic conditions such as cervical intraepithelial neoplasia are admissible.
* Endocrine disease including thyroid disease (recently diagnosed or whose medication dose is not stable), adrenal disease, diabetes mellitus (pregestational and gestational).
* Renal disease with altered renal function (creatinine > 0.9, proteinuria > 300 mg/24 hour)
* Epilepsy or other seizure disorder
* Any collagen disease (lupus erythematosus, scleroderma, etc.)
* Active liver disease (acute hepatitis, chronic active hepatitis, persistently abnormal liver enzymes). Liver disorders accounting for cholestasis (including cholestasis of pregnancy) if diagnosed prior to enrollment.
* Hematological disorder including alloimmune and isoimmune thrombocytopenia but excluding mild iron deficiency anemia (Hb > 9 gm/dl). Patients with sickle cell disease are excluded.
* Chronic pulmonary disease including asthma requiring regular use of medication and active TB. An asthma inhaler used on an as needed basis for a cold or an asthma attack is not considered regular use.
* Heart disease except mitral value prolapse not requiring medication
* Cardiovascular disorders: chronic hypertension, gestational hypertension or preeclampsia diagnosed prior to enrollment
* Infectious diseases: HIV, CMV, toxoplasmosis, parvovirus B19, HBV, HCV
* Chronic treatments with medications such as aspirin, steroids, anti-hypertensive agents, immunosuppressants, antineoplastic drugs.
* Prior laparoscopic or open uterine surgeries where the uterine cavity was entered (such as myomectomies)
* Resectoscopic myomectomies (prior resectoscopic polypectomies are not contraindications)
* Prior classical cesarean deliveries.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study enrolls low risk pregnant women
Enrollment: 1566 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Number of prenatally identified fetuses that will be classified as small or large for gestational age as infants (SGA and LGA infants) | From enrollment through study completion, an average of 1 year. Prenatal evaluation of fetal growth and amniotic fluid volume will be performed at 35-38, 40,41, and 41+ weeks' gestation. Infants' weights will be evaluated at birth
  Birthweight percentile will be classified according to the INeS neonatal charts (Bertino 2010) to identify SGA (birthweight < 10th percentile) , LGA (birthweight > 90th percentile) and AGA (appropriate for gestational age, whose birthweight ranges between the 10th and the 90th percentile) infants.

SECONDARY OUTCOMES:
Number of formal obstetric ultrasound (US) requested due to abnormal fetal growth or amniotic fluid suspected prenatally | From enrollment through study completion, an average of 1 year. Formal obstetric ultrasound will be requested in case of suspicion of abnormal fetal growth or amniotic fluid on screening with symphysis fundal height associated or not to POC ultrasound
  Formal obstetric ultrasound are the ones performed by trained perinatologists in the prenatal diagnosis department
Number of cases of oligohydramnios and polyhydramnios identified on formal obstetric US after being suspected on prenatal evaluation | From enrollment through study completion, an average of 1 year. Formal obstetric ultrasound will be requested in case of suspicion of abnormal fetal growth or amniotic fluid on screening with symphysis fundal height associated or not to POC ultrasound
  Formal obstetric ultrasound are the ones performed by trained perinatologists in the prenatal diagnosis department
Number of deliveries indicated by amniotic fluid or fetal growth abnormalities detected on formal obstetric US | At the time of delivery, from enrollment through study completion, an average of 1 year
  Indicated deliveries are inductions of labor or cesarean deliveries performed in non-laboring women due to amniotic fluid or fetal growth abnormalities
Number of adverse neonatal outcome cases | At the time of delivery, from enrollment through study completion, an average of 1 year
  Adverse neonatal outcomes are summarized as a composite of neonatal death, non-invasive (cPAP) or invasive (mechanical ventilation) respiratory support, hypoglycemia (< 44 mg/dl needing therapy), newborn sepsis, confirmed seizures, stroke, intraventricular hemorrhage (IVH), basal nuclei anomalies, cardiopulmonary resuscitation, umbilical-cord-blood arterial pH < 7.0 or base excess < -12.5, prolonged hospitalization (> 5 days), or shoulder dystocia
Number of adverse maternal outcome cases | At the time of delivery, from enrollment through study completion, an average of 1 year
  Adverse maternal outcomes are summarized as a composite of blood loss > 1000 ml, maternal sepsis, post-partum endometritis, hysterectomy, bowel or urinary tract injuries, uterine rupture, wound (either perineal or abdominal) complications (i.e abscess, hematoma or disruption), 3rd and 4th degree perineal lacerations, blood transfusion, maternal admission to the ICU, laparotomy, and death

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Chiossi, MD, Principal Investigator — University of Modena and Reggio Emilia, Modena Policlinico Hospital, Department of Obstetrics and Gynecology
Locations (3):
- Italy (3):
  - Azienda Ospedaliero Universitaria Policlinico di Modena, Modena, Modena
  - Cesena Hospital, Cesena
  - Foundation MBBM at San Gerardo Hospital, University of Milan-Bicocca School of Medicine and Surgery, Monza, Italy., Monza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Hafez L, Chauhan SP, Riegel M, Balogun OA, Hammad IA, Berghella V. Routine third-trimester ultrasound in low-risk pregnancies and perinatal death: a systematic review and meta-analysis. Am J Obstet Gynecol MFM. 2020 Nov;2(4):100242. doi: 10.1016/j.ajogmf.2020.100242. Epub 2020 Oct 3. PMID 33345941
- [Background] Committee on Practice Bulletins-Obstetrics and the American Institute of Ultrasound in Medicine. Practice Bulletin No. 175: Ultrasound in Pregnancy. Obstet Gynecol. 2016 Dec;128(6):e241-e256. doi: 10.1097/AOG.0000000000001815. No abstract available. PMID 27875472
- [Background] Macrosomia: ACOG Practice Bulletin, Number 216. Obstet Gynecol. 2020 Jan;135(1):e18-e35. doi: 10.1097/AOG.0000000000003606. PMID 31856124
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics and the Society forMaternal-FetalMedicin. ACOG Practice Bulletin No. 204: Fetal Growth Restriction. Obstet Gynecol. 2019 Feb;133(2):e97-e109. doi: 10.1097/AOG.0000000000003070. PMID 30681542
- [Background] Bertino E, Spada E, Occhi L, Coscia A, Giuliani F, Gagliardi L, Gilli G, Bona G, Fabris C, De Curtis M, Milani S. Neonatal anthropometric charts: the Italian neonatal study compared with other European studies. J Pediatr Gastroenterol Nutr. 2010 Sep;51(3):353-61. doi: 10.1097/MPG.0b013e3181da213e. PMID 20601901
- [Background] Blue NR, Yordan JMP, Holbrook BD, Nirgudkar PA, Mozurkewich EL. Abdominal Circumference Alone versus Estimated Fetal Weight after 24 Weeks to Predict Small or Large for Gestational Age at Birth: A Meta-Analysis. Am J Perinatol. 2017 Sep;34(11):1115-1124. doi: 10.1055/s-0037-1604059. Epub 2017 Jul 3. No abstract available. PMID 28672412
- [Background] Bricker L, Medley N, Pratt JJ. Routine ultrasound in late pregnancy (after 24 weeks' gestation). Cochrane Database Syst Rev. 2015 Jun 29;2015(6):CD001451. doi: 10.1002/14651858.CD001451.pub4. PMID 26121659
- [Background] Caradeux J, Martinez-Portilla RJ, Peguero A, Sotiriadis A, Figueras F. Diagnostic performance of third-trimester ultrasound for the prediction of late-onset fetal growth restriction: a systematic review and meta-analysis. Am J Obstet Gynecol. 2019 May;220(5):449-459.e19. doi: 10.1016/j.ajog.2018.09.043. Epub 2019 Jan 8. PMID 30633918
- [Background] Chauhan SP, Cole J, Sanderson M, Magann EF, Scardo JA. Suspicion of intrauterine growth restriction: Use of abdominal circumference alone or estimated fetal weight below 10%. J Matern Fetal Neonatal Med. 2006 Sep;19(9):557-62. doi: 10.1080/14767050600798267. PMID 16966124
- [Background] Doyle LW. Long-term neurologic outcome for the very preterm growth-restricted fetus. Pediatrics. 2011 Apr;127(4):e1048-9. doi: 10.1542/peds.2011-0262. Epub 2011 Mar 7. No abstract available. PMID 21382952
- [Background] Society for Maternal-Fetal Medicine (SMFM). Electronic address: pubs@smfm.org; Martins JG, Biggio JR, Abuhamad A. Society for Maternal-Fetal Medicine Consult Series #52: Diagnosis and management of fetal growth restriction: (Replaces Clinical Guideline Number 3, April 2012). Am J Obstet Gynecol. 2020 Oct;223(4):B2-B17. doi: 10.1016/j.ajog.2020.05.010. Epub 2020 May 12. PMID 32407785
- [Background] Goto E. Symphysis-fundal height to identify large-for-gestational-age and macrosomia: a meta-analysis. J Obstet Gynaecol. 2020 Oct;40(7):929-935. doi: 10.1080/01443615.2019.1673713. Epub 2019 Dec 8. PMID 31814480
- [Background] Henrichs J, Verfaille V, Jellema P, Viester L, Pajkrt E, Wilschut J, van der Horst HE, Franx A, de Jonge A; IRIS study group. Effectiveness of routine third trimester ultrasonography to reduce adverse perinatal outcomes in low risk pregnancy (the IRIS study): nationwide, pragmatic, multicentre, stepped wedge cluster randomised trial. BMJ. 2019 Oct 15;367:l5517. doi: 10.1136/bmj.l5517. PMID 31615781
- [Background] Lees CC, Stampalija T, Baschat A, da Silva Costa F, Ferrazzi E, Figueras F, Hecher K, Kingdom J, Poon LC, Salomon LJ, Unterscheider J. ISUOG Practice Guidelines: diagnosis and management of small-for-gestational-age fetus and fetal growth restriction. Ultrasound Obstet Gynecol. 2020 Aug;56(2):298-312. doi: 10.1002/uog.22134. No abstract available. PMID 32738107
- [Background] Lindhard A, Nielsen PV, Mouritsen LA, Zachariassen A, Sorensen HU, Roseno H. The implications of introducing the symphyseal-fundal height-measurement. A prospective randomized controlled trial. Br J Obstet Gynaecol. 1990 Aug;97(8):675-80. doi: 10.1111/j.1471-0528.1990.tb16237.x. PMID 2205286
- [Background] Lindqvist PG, Molin J. Does antenatal identification of small-for-gestational age fetuses significantly improve their outcome? Ultrasound Obstet Gynecol. 2005 Mar;25(3):258-64. doi: 10.1002/uog.1806. PMID 15717289
- [Background] Nicolini U, Todros T, Ferrazzi E, Zorzoli A, Groli C, Zucca S, Tinti A, Dodero D, Destro F, Ceccarello P, et al. [Transverse fetal growth curves. A multicenter study]. Minerva Ginecol. 1986 Nov;38(11):873-87. No abstract available. Italian. PMID 3808422
- [Background] Moraitis AA, Shreeve N, Sovio U, Brocklehurst P, Heazell AEP, Thornton JG, Robson SC, Papageorghiou A, Smith GC. Universal third-trimester ultrasonic screening using fetal macrosomia in the prediction of adverse perinatal outcome: A systematic review and meta-analysis of diagnostic test accuracy. PLoS Med. 2020 Oct 13;17(10):e1003190. doi: 10.1371/journal.pmed.1003190. eCollection 2020 Oct. PMID 33048935
- [Background] Papageorghiou AT, Ohuma EO, Gravett MG, Hirst J, da Silveira MF, Lambert A, Carvalho M, Jaffer YA, Altman DG, Noble JA, Bertino E, Purwar M, Pang R, Cheikh Ismail L, Victora C, Bhutta ZA, Kennedy SH, Villar J; International Fetal and Newborn Growth Consortium for the 21st Century (INTERGROWTH-21st). International standards for symphysis-fundal height based on serial measurements from the Fetal Growth Longitudinal Study of the INTERGROWTH-21st Project: prospective cohort study in eight countries. BMJ. 2016 Nov 7;355:i5662. doi: 10.1136/bmj.i5662. PMID 27821614
- [Background] Pay AS, Wiik J, Backe B, Jacobsson B, Strandell A, Klovning A. Symphysis-fundus height measurement to predict small-for-gestational-age status at birth: a systematic review. BMC Pregnancy Childbirth. 2015 Feb 10;15:22. doi: 10.1186/s12884-015-0461-z. PMID 25884884
- [Background] Robert Peter J, Ho JJ, Valliapan J, Sivasangari S. Symphysial fundal height (SFH) measurement in pregnancy for detecting abnormal fetal growth. Cochrane Database Syst Rev. 2015 Sep 8;2015(9):CD008136. doi: 10.1002/14651858.CD008136.pub3. PMID 26346107
- [Background] Sovio U, White IR, Dacey A, Pasupathy D, Smith GCS. Screening for fetal growth restriction with universal third trimester ultrasonography in nulliparous women in the Pregnancy Outcome Prediction (POP) study: a prospective cohort study. Lancet. 2015 Nov 21;386(10008):2089-2097. doi: 10.1016/S0140-6736(15)00131-2. Epub 2015 Sep 7. PMID 26360240
- [Background] Sparks TN, Cheng YW, McLaughlin B, Esakoff TF, Caughey AB. Fundal height: a useful screening tool for fetal growth? J Matern Fetal Neonatal Med. 2011 May;24(5):708-12. doi: 10.3109/14767058.2010.516285. Epub 2010 Sep 17. PMID 20849205
- [Background] von Beckerath AK, Kollmann M, Rotky-Fast C, Karpf E, Lang U, Klaritsch P. Perinatal complications and long-term neurodevelopmental outcome of infants with intrauterine growth restriction. Am J Obstet Gynecol. 2013 Feb;208(2):130.e1-6. doi: 10.1016/j.ajog.2012.11.014. Epub 2012 Nov 15. PMID 23159694
- See also: NICE. Antenatal care for uncomplicated pregnancies. 2008. — http://www.nice.org.uk/guidance/cg62/chapter/guidance.